CLINICAL TRIAL: NCT03570554
Title: A Pilot Study Assessing the Treatment Responsiveness of a Novel Osteoarthritis Stiffness Scale
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19783
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Naproxen; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A-D-C-B (Experimental): Participants received naproxen 660 mg daily for 3 days and 440 mg on the fourth day; followed by placebo for 4 days; followed by celecoxib 200 mg daily for 3 days and 100 mg on the fourth day; followed by acetaminophen 3900 mg daily for 3 days and 1300 mg on the fourth day. Treatment periods were separated by a washout period of 3 to 7 days.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetaminophen ER; Drug: Celecoxib; Drug: Placebo
- Treatment B-C-D-A (Experimental): Participants received acetaminophen 3900 mg daily for 3 days and 1300 mg on the fourth day; followed by celecoxib 200 mg daily for 3 days and 100 mg on the fourth day; followed by placebo for 4 days; followed by naproxen 660 mg daily for 3 days and 440 mg on the fourth day. Treatment periods were separated by a washout period of 3 to 7 days.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetaminophen ER; Drug: Celecoxib; Drug: Placebo
- Treatment C-A-B-D (Experimental): Participants received celecoxib 200 mg daily for 3 days and 100 mg on the fourth day; followed by naproxen 660 mg daily for 3 days and 440 mg on the fourth day; followed by acetaminophen 3900 mg daily for 3 days and 1300 mg on the fourth day; followed by placebo for 4 days. Treatment periods were separated by a washout period of 3 to 7 days.
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetaminophen ER; Drug: Celecoxib; Drug: Placebo
- Treatment D-B-A-C (Experimental): Participants received placebo for 4 days; followed by acetaminophen 3900 mg daily for 3 days and 1300 mg on the fourth day; followed by naproxen 660 mg daily for 3 days and 440 mg on the fourth day; followed by celecoxib 200 mg daily for 3 days and 100 mg on the fourth day. Treatment periods were separated by a washout period of 3 to 7 days
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031); Drug: Acetaminophen ER; Drug: Celecoxib; Drug: Placebo

INTERVENTIONS:
Drug: Naproxen Sodium (Aleve, BAY117031) — 660 mg daily for 3 days, 440 mg on the fourth day, over-encapsulated tablet, oral (Treatment A)
Drug: Acetaminophen ER — 3900 mg daily for 3 days, 1300 mg on the fourth day, over-encapsulated extended release (ER) tablet, oral (Treatment B)
Drug: Celecoxib — 200 mg daily for 3 days, 100 mg on the fourth day, over-encapsulated capsule, oral (Treatment C)
Drug: Placebo — Over-encapsulation capsule, 4 days, oral (Treatment D)

SUMMARY:
Osteoarthritis is a common, chronic, progressive, skeletal, degenerative disorder that frequently affects several joints such as knee, hip, spine and hands.This placebo-controlled clinical trial assessed the effects of naproxen sodium, acetaminophen and celecoxib on stiffness in subjects with osteoarthritis.

DETAILED DESCRIPTION:
The primary objective of the study was to assess the responsiveness of the Brief Arthritis Stiffness Scale (BASS) for detecting treatment effects of common over-the-counter (OTC) analgesics and a common prescription analgesic in subjects with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years
* Body Mass Index (BMI) between 18 and <40 kg/m^2
* Unilateral or bilateral osteoarthritis of the knee
* Diagnostic quality radiography of the target knee performed no more than 1 year prior to baseline showing evidence of osteoarthritis (OA) with Kellgren and Lawrence grade of II or III
* Joint Stiffness Severity score ≥3.0 on a 0-10 numerical rating scale (NRS) at screening

Exclusion Criteria:

* History of underlying inflammatory arthropathy, rheumatoid arthritis or fibromyalgia
* History of or scheduled for target knee replacement surgery
* Recent injury in target knee (past 4 months)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Radiant Research, Inc., Chandler, Arizona
  - Radiant Research, Inc., Pinellas Park, Florida
  - Radiant Research, Inc., Chicago, Illinois
  - Radiant Research, Inc., Cincinnati, Ohio
  - Radiant Research, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in the US between 29 June 2018 (first participant first visit) and 14 June 2019 (last participant last visit).
Pre-assignment Details: Overall, 209 participants were screened. Of them, 168 participants were screen failures, and 41 subjects were randomized to study treatments.
Period: Overall Study
Arm/Group | Treatment A-D-C-B | Treatment B-C-D-A | Treatment C-A-B-D | Treatment D-B-A-C
Started | 10 | 10 | 11 | 10
Completed | 10 | 10 | 10 | 9
Not Completed | 0 | 0 | 1 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least one dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A-D-C-B | Treatment B-C-D-A | Treatment C-A-B-D | Treatment D-B-A-C | Total
Number analyzed (Participants) | 10 | 10 | 11 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (9.20) | 61.3 (8.77) | 61.6 (7.55) | 59.6 (8.28) | 61.2 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 11 | 7 | 33
  Male | 1 | 4 | 0 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 4
  Not Hispanic or Latino | 9 | 10 | 9 | 9 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 2 | 5 | 16
  White | 6 | 5 | 8 | 5 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Brief Arthritis Stiffness Scale (BASS) [Mean (Standard Deviation); unit: Scores on a scale] — Brief Arthritis Stiffness Scale (BASS) is a patient-reported outcome (PRO) instrument measuring of the severity of osteoarthritis-related stiffness in the target knee joint. The BASS score ranges from 0 to 40 and a higher score indicates worse stiffness. Population: Participants in safety population with evaluable data for this characteristic
  Scores on a scale
    Treatment period 1: number analyzed (Participants) | 10 | 10 | 11 | 9 | 40
    Treatment period 1 | 26.7 (4.90) | 25.8 (5.05) | 27.8 (5.56) | 23.1 (5.35) | 26.0 (5.31)
    Treatment period 2: number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
    Treatment period 2 | 25.8 (7.74) | 21.8 (8.32) | 22.3 (9.74) | 25.3 (4.64) | 23.8 (7.74)
    Treatment period 3: number analyzed (Participants) | 10 | 10 | 10 | 9 | 39
    Treatment period 3 | 26.3 (5.56) | 17.7 (10.03) | 22.9 (10.29) | 24.0 (6.48) | 22.7 (8.69)
    Treatment period 4: number analyzed (Participants) | 10 | 10 | 10 | 9 | 39
    Treatment period 4 | 21.9 (10.56) | 20.3 (6.40) | 24.2 (9.95) | 23.8 (7.92) | 22.5 (8.68)

OUTCOME MEASURES:

1. Primary Outcome: Sum of Change in Brief Arthritis Stiffness Scale (BASS) Scores Over the 4-day Treatment Period
Description: Brief Arthritis Stiffness Scale (BASS) is a patient-reported outcome (PRO) instrument measuring of the severity of osteoarthritis-related stiffness in the target knee joint. The BASS score ranges from 0 to 40 and a higher score indicates worse stiffness. This endpoint was calculated by summing the changes from baseline (CFB) in BASS scores at Days 2, 3, and 4 of the treatment periods.
Time Frame: 4 days
Population: Per-protocol (PP) population: all subjects who were randomly assigned and had taken at least one dose of IMP without major protocol violations that could affect the evaluability of the primary efficacy parameter.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Groups:
- Naproxen: Participants received naproxen 660 mg daily for 3 days and 440 mg on the fourth day.
- Acetaminophen ER: Participants received acetaminophen 3900 mg daily for 3 days and 1300 mg on the fourth day.
- Celecoxib: Participants received celecoxib 200 mg daily for 3 days and 100 mg on the fourth day.
- Placebo: Participants received placebo for 4 days.
Arm/Group | Naproxen | Acetaminophen ER | Celecoxib | Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 36
Scores on a scale | -12.6 (5.46) | -13.6 (5.46) | -11.7 (5.46) | -2.3 (5.47)

2. Secondary Outcome: Absolute Brief Arthritis Stiffness Scale (BASS) Score at Each Time Point
Description: Brief Arthritis Stiffness Scale (BASS) is a patient-reported outcome (PRO) instrument measuring of the severity of osteoarthritis-related stiffness in the target knee joint. The BASS score ranges from 0 to 40 and a higher score indicates worse stiffness.
Time Frame: 4 days
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Naproxen | Acetaminophen ER | Celecoxib | Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 36
Scores on a scale
  Day 1 | 23.0 (1.84) | 23.3 (1.84) | 24.6 (1.84) | 22.6 (1.85)
  Day 2 | 20.8 (1.62) | 19.7 (1.62) | 20.6 (1.62) | 23.2 (1.62)
  Day 3 | 18.4 (1.97) | 18.4 (1.97) | 18.9 (1.98) | 22.4 (1.98)
  Day 4 | 18.1 (1.97) | 18.0 (1.97) | 18.5 (1.97) | 22.0 (1.97)

3. Secondary Outcome: Change From Baseline in Brief Arthritis Stiffness Scale (BASS) Score at Day 4
Description: as for outcome 2
Time Frame: Day 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Naproxen | Acetaminophen ER | Celecoxib | Placebo
Number analyzed (Participants) | 37 | 37 | 37 | 36
Scores on a scale | -5.2 (1.97) | -5.3 (1.97) | -4.8 (1.97) | -1.3 (1.97)

ADVERSE EVENTS:
Time Frame: After the first dose of the investigational medicinal product (IMP) until the end of the treatment phase, up to 37 days
Arm/Group | Naproxen | Acetaminophen ER | Celecoxib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40 | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 5/39 | 8/40 | 10/40 | 3/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen (N=39) | Acetaminophen ER (N=40) | Celecoxib (N=40) | Placebo (N=39)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT03570554/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT03570554/SAP_001.pdf